CLINICAL TRIAL: NCT01132144
Title: Endometrial Injury Prior Ovulation Induction for Assisted Reproductive Techniques: a Randomized Controlled Trial
Brief Title: Endometrial Injury for Assisted Reproduction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped after safety analysis because of significant benefit of intervention.
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Apoio ao Ensino, Pesquisa e Assistência do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Wellington P Martins, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCRP10340/09
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Infertility
Keywords: Reproductive Techniques; Embryo Implantation; Endometrium; Ultrasonography
MeSH Terms: conditions — Infertility | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endometrial injury group (Experimental): Endometrial biopsy was performed once with a pipelle de Cornier® in the month before initiating controlled ovarian stimulation.
  Interventions: Procedure: Endometrial injury
- Control group (Sham Comparator): Introduction of the speculum and wiping of the cervix with gaze for 30 seconds.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Endometrial injury — Evaluate the position and size of the uterus by transabdominal ultrasonography, with the bladder comfortably full.
  Identify the cervix with a disposable speculum. Open one sealed opaque envelope for allocation.
  Endometrial injury:
  * Slide the Pipelle de Cornier® (Laboratoires Prodimed, Neully-En-Thelle, France) gently through the cervix up to the uterine fundus. Transbadominal ultrasound might be used to confirm position.
  * Draw back the piston to the end of the biopsy cannula until it locks creating a negative pressure.
  * Sweep the uterine fundus slowly several times up to the internal orifice of the cervix, using regular to-and-fro movements while rotating the sampler to include the whole uterine cavity in the specimen, for 30 seconds or until participant ask for stopping.
  Arms: Endometrial injury group
Procedure: Control group — The investigator will dry the cervix with gauze and forceps for for 30 seconds or until participant ask for stopping.
  Other Names: Sham procedure
  Arms: Control group

SUMMARY:
The objective of this study is to evaluate the effect of endometrial injury performed prior ovulation induction for assisted reproductive techniques main outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women who will start assisted reproductive techniques with planned fresh embryo transfer.
* Age between 18 and 38 years.
* Written informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wellington P Martins, PhD, Principal Investigator — Faculdade de Medicina de Ribeirão Preto, Universidade de São Paulo
Locations (1):
- Setor de Reproducao Humana do HC-FMRP-USP, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Lensen SF, Armstrong S, Gibreel A, Nastri CO, Raine-Fenning N, Martins WP. Endometrial injury in women undergoing in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Jun 10;6(6):CD009517. doi: 10.1002/14651858.CD009517.pub4. PMID 34110001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment occurred from July 2010 to March 2012 in the fertility clinic of an university hospital.
Pre-assignment Details: All women that fulfilled eligibility criteria were invited to participate. Those who agreed were included. No women was excluded.
Groups:
- Endometrial Injury Group: Endometrial biopsy was performed once with a pipelle de Cornier® in the month before initiating controlled ovarian stimulation. The pipelle was introduced gently through the cervix up to the uterine fundus. The piston was then drawn back to the end of the biopsy cannula until it self-locks and creates a negative pressure. Aiming to wound the entire endometrium, the examiner applied regular back-and-forth movements while rotating the sampler covering the whole uterine cavity. This procedure was continued until fragments of uterine mucosa appeared within the sheath, which generally took 30 seconds.
Period: Overall Study
Arm/Group | Endometrial Injury Group | Control Group
Started | 79 | 79
Completed | 79 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometrial Injury Group | Control Group | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 79 | 79 | 158
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (3.2) | 32.1 (3.1) | 32.2 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 79 | 158
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 79 | 79 | 158

OUTCOME MEASURES:

1. Primary Outcome: Live Birth
Description: The complete expulsion or extraction from its mother of a product of fertilization, irrespective of the duration of the pregnancy, which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation, or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached.
  Note: All allocated women will be used as denominator when assessing live birth rate.
Time Frame: 1 year
Population: All women enrolled.
Measure: Number; unit: participants
Arm/Group | Endometrial Injury Group | Control Group
Number analyzed (Participants) | 79 | 79
participants | 33 | 18

2. Secondary Outcome: Clinical Pregnancy
Description: Pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy. Multiple gestational sacs are counted as one clinical pregnancy.
  Note: All allocated women will be considered when assessing clinical pregnancy rate.
Time Frame: 3 months
Population: All women enrolled.
Measure: Number; unit: participants
Arm/Group | Endometrial Injury Group | Control Group
Number analyzed (Participants) | 79 | 79
participants | 39 | 23

3. Secondary Outcome: Ongoing Pregnancy
Description: At least one fetus with heart beat after 12 weeks of gestational age.
  Note: All allocated women will be considered when assessing ongoing pregnancy rate.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Endometrial Injury Group | Control Group
Number analyzed (Participants) | 79 | 79
participants | 33 | 18

4. Secondary Outcome: Miscarriage
Description: Loss of a clinical pregnancy before 20 completed weeks of gestational age (18 weeks after fertilization).
  Note: All allocated women will be considered when assessing miscarriage rate.
Time Frame: 9 months
Population: The number of clinical pregnancies was used as denominator, since miscarriage is a harm that can only happen in pregnant women.
Measure: Number; unit: Clinical pregnancies
Arm/Group | Endometrial Injury Group | Control Group
Number analyzed (Participants) | 39 | 23
Clinical pregnancies | 6 | 5

5. Secondary Outcome: Implantation Rate
Description: The number of gestational sacs observed divided by the number of embryos transferred.
Time Frame: 3 months
Reporting Status: Not Posted

6. Secondary Outcome: Endometrial Thickness
Description: The maximum distance perpendicular to the inter-endometrial interface from the endometrium-myometrium interface of the anterior to the posterior wall of the uterus assessed in the sagittal plane. This outcome will be assessed when at least one follicle ≥ 17mm is observed.
Time Frame: 1 month
Population: Women that achieved at least one follicle >17mm during ovarian stimulation.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Endometrial Injury Group | Control Group
Number analyzed (Participants) | 72 | 74
mm | 10.12 (1.55) | 9.98 (1.62)

7. Secondary Outcome: Endometrial Volume
Description: The total volume of endometrial tissue assessed by three-dimensional ultrasonography. This outcome will be assessed when at least one follicle ≥ 17mm is observed.
Time Frame: 1 month
Population: Women that achieved at least one follicle >17mm during ovarian stimulation.
Measure: Mean (Standard Deviation); unit: cm³
Arm/Group | Endometrial Injury Group | Control Group
Number analyzed (Participants) | 72 | 74
cm³ | 6.18 (1.63) | 6.01 (1.48)

8. Secondary Outcome: Three-dimensional Doppler Indices From Endometrium (VFI)
Description: Vascularization index (VI), flow index (FI) and vascularization-flow index (VFI) assessed from endometrium using three-dimensional Power Doppler ultrasonography. This outcome will be assessed when at least one follicle ≥ 17mm is observed.
  Only VFI was reported as it is a combination of VI and FI (VFI = VI*FI/100), and currently there are several concerns about the validity of these indices.
  Such indices have no scale.
Time Frame: 1 month
Population: Women that achieved at least one follicle >17mm during ovarian stimulation.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Endometrial Injury Group | Control Group
Number analyzed (Participants) | 72 | 74
index | 0.97 (0.51) | 0.76 (0.40)

9. Secondary Outcome: Procedure Related Pain
Description: Pain will be assessed using a Visual Analogue Scale (VAS). We will use a 10 cm length horizontal line, anchored by word descriptors at each end: "No Pain" = 0 cm and "Very Severe Pain" = 10 cm.
  This outcome will be assessed in both groups, just after endometrial injury or sham procedure.
Time Frame: Immediately after procedure
Population: All women enrolled.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Endometrial Injury Group | Control Group
Number analyzed (Participants) | 79 | 79
cm | 6.42 (2.35) | 1.82 (1.52)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Major fetal malformation. The occurrence of major fetal malformation detected at birth was assessed by phone interview with the parents.
Arm/Group | Endometrial Injury Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/79
Other Adverse Events (participants affected / at risk) | 0/79 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No